CLINICAL TRIAL: NCT06675734
Title: Pain Management After Free Gingival Graft Surgery: Effectiveness of Different Analgesic Strategies
Brief Title: Pain Management After Free Gingival Graft Surgery
Status: Completed | Type: Observational
Sponsor: Istanbul Aydın University (Other)
Responsible Party: Principal Investigator, Ezgi Sıla Taşkaldıran, IstanbulAU, Istanbul Aydın University
Other Study IDs: 2023/148
Record Dates: First submitted 2024-11-04; First posted 2024-11-05 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Gingival Recession, Localized; Gingival Recession, Generalized; Gingival Recession, Mucogingival Surgery
Keywords: free gingival graft; pain management; PROM; gingival augmentation
MeSH Terms: conditions — Gingival Recession; Agnosia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Experimental Group (Group E): After the operation, study groups will be formed according to the post operative analgesia method determined and applied by the periodontologist. Accordingly, individuals to whom diclofenac sodium-containing ampoule was administered intramuscularly within 1 hour following the operation will be included in the study group.
  Interventions: Drug: diclofenac sodium solution
- Control Group (Group C): Patients who do not require intramuscular administration of diclofenac sodium containing ampoule will be included in the control group.

INTERVENTIONS:
Drug: diclofenac sodium solution — The experimental group consisted of patients in whom diclofenac sodium was administered IM and the control group consisted of patients in whom diclofenac sodium was administered orally only.
  Groups: Experimental Group (Group E)

SUMMARY:
Keratinized gingiva reduces the risk of gingival disease and infection by protecting the tissue around the teeth and is therefore very important for gingival health. Free gingival grafting is a widely used technique in periodontal surgery. It is used to correct gum recession or to support the tissue around dental implants. Free gingival grafting involves taking the patient's own gum tissue from another area and transplanting it to the area in need. This method is an effective way to restore periodontal health and achieve esthetic results. Scientific studies show that free gum grafting is successful in treating gum recession and preventing complications from implant surgery. However, as with all surgical procedures, several complications can occur after free gum surgery. The most prominent of these is postoperative pain. Although various methods of pain prevention have been proposed in the literature, the most appropriate pain management strategy has not been described. The aim of this study was to evaluate the effect of analgesia methods on postoperative pain level after free gingival grafting.

DETAILED DESCRIPTION:
Human keratinized gingiva includes free and adherent gingival portions and extends from the gingival margin to the mucogingival junction. Clinical studies have concluded that a keratinized gingival margin of at least 2 mm in width is required to maintain periodontal health around teeth. Similar to periodontal health, it has been reported that insufficient keratinized gingival width in the peri-implant region can lead to problems such as plaque accumulation, pain during brushing, increased gingival inflammation, gingival recession and peri-implant bone loss. To avoid all these problems, a number of surgical procedures have been proposed to increase the width of the keratinized gingiva. Among the surgical procedures used to increase the width of the keratinized gingiva, free gingival grafting stands out for its ease of use and the fact that it requires no additional material. Free gingival grafting is an effective way to restore periodontal health and achieve esthetic results. Scientific studies show that free gingival grafting is a successful method for treating gingival recession and preventing complications in implant surgery.In free gingival grafting, the epithelial graft from the palate leaves an open wound surface that can take 2 to 4 weeks to heal. Accordingly, the most common postoperative problem is pain at the recipient and donor sites. Various surgical techniques and a number of postoperative applications have been proposed in the literature to prevent pain. These studies have mostly focused on pain control at the donor site. For example, in a study conducted with the hypothesis that an epithelial graft harvested from the donor site in a smaller size compared to traditional methods may cause less pain, it was reported that graft size had no effect on postoperative pain. On the other hand, the efficacy of different applications on the palatal wound area after free gingival transplantation using the traditional method has also been evaluated. In a systematic review, platelet-rich fibrin membrane applied to protect the donor site after surgery was shown to reduce the pain symptom. In a randomized controlled trial, a low-dose laser was also applied to the donor site, and it was reported that postoperative pain was less than in individuals without laser application. Although there are studies evaluating donor site pain control after free gingival surgery, there is no study evaluating the patient's pain control systemically. Our study was designed to contribute to the literature in this regard.

ELIGIBILITY:
Inclusion Criteria:

* individuals who underwent a free gingival graft operation in which the donor site was used as the palatinal region

Exclusion Criteria:

* pre-operative and post-operative complications
* The presence of any condition that prevents reading and understanding,
* Being unable to comply with the control sessions,
* Being on psychiatric medication.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Individuals who underwent free gingival surgery in the clinics of Istanbul Aydın University Faculty of Dentistry, Department of Periodontology.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2023-11-29 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-05-27 (Actual)

PRIMARY OUTCOMES:
VAS | 7 days post-operatively
  Post-operative VAS Pain Scale
Medication | 7 days post-operatively
  Amount of post-operative pain medication use

SECONDARY OUTCOMES:
PROMs | 3 days post-operatively
  Patient-reported outcome measures questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Ezgi Sila Taskaldiran, PhD, Study Director — Istanbul Aydın University
Locations (1):
- Istanbul Aydin University Dentistry Faculty, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No